CLINICAL TRIAL: NCT03193489
Title: A High-intensity Multi-component Agility Intervention in Parkinson's Patients: Two-year Follow-up
Brief Title: Two-year Follow-up to High-intensity Multi-component Agility Intervention That Improves Clinical and Motor Symptoms of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Tollár József, Principal investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKEB0013/2015
Record Dates: First submitted 2017-06-01; First posted 2017-06-20 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2017-06

CONDITIONS: Follow up; Parkinson Disease; Rehabilitation
Keywords: Balance; Posturograpy; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise therapy (Experimental): Parkinson's group takes part in a treadmill treatment that takes place 3 times a week for 2 years.
  Interventions: Other: Follow-up; Other: Post-treatment control; Other: Control Parkinson group

INTERVENTIONS:
Other: Follow-up
Other: Post-treatment control — After 3 weeks of intensive treatment, no special exercises are performed as a control.
Other: Control Parkinson group — No treatment.

SUMMARY:
Individualization of exercise is recommended but rarely performed in patients with Parkinson's disease (PD).

Unusually High Intensity and Individual Sensor Motor with Visuomotor Mobility Trainer The clinical symptoms, mobility and posture of PD patients. After 3 weeks of intensive treatment, treated patients and the control group were subjected to a two-year observation.

Objectives: The effect of the unusually highly intense and strictly individualized sensomotor and visuomotor agility program was determined for the clinical symptoms, mobility and stability of non-demented PD patients with a two-year follow-up. Detection and comparison of results of patients undergoing biphasic maintenance with the results of intensively treated patients and the control group.

Patients were recalled every 3 months after the first intensive examination and one year after a one-year control. The results of the active group were continuously compared with the results of the passive and control groups, thus determining the effectiveness of our treatment and the deterioration of the other groups in life-quality.

The treated groups will be divided into two. One Parkinson's group takes part in a treadmill treatment that takes place 3 times a week for 2 years. The other group does not undergo a special series of exercises after 3 weeks of intensive therapy.

Main outcome measures: Movement disorder Society Unified Parkinson Disease Rating Scale, Motor Experiences of Daily Living, a measure sensitive to changes in a broad spectrum of PD symptoms.

In group time, repeated measurements of variance analysis were compared to MDS-UPDRS M-EDL, Beck Depression Score, PDQ-39, EQ5D VAS, Schwab & England Scale for Parkinson's Disease. The TUG test and 12 static posturographic measurements are compared and compared to the healthy group as a standard.

An at-limit and individualized sensorimotor and visuomotor agility exercise program vs. standard care, will improve non-demeted, stage 2-3 PD patient's clinical symptoms, mobility, and postural stability by functionally meaningful margins. As a long-term solution, a follow-up treatment can slow down the progression of clinical symtoms.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Hoenh Yahr scale of 2-3
* Instability problem

Exclusion Criteria:

* Severe heart problems
* Severe demeanor
* Alcoholism
* Drug problems

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L | 0-5 scale (2 year-long, higher point is better)
  Questionnaire
posturography | mm (2 year-long, the smaller the mm the better the result)
  body sway, Objective measurement of holding instability
Timed up and Go test | sec (2 year-long, the less time you take the test, the better the result )
  Measuring the speed of walking

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Related Info — https://www.ncbi.nlm.nih.gov/pubmed/